CLINICAL TRIAL: NCT05506384
Title: Treatment Study for Problematic Gaming and Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-04797
Record Dates: First submitted 2022-08-08; First posted 2022-08-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Pathological Gambling; Internet Gaming Disorder
Keywords: Gaming; Gambling; Adolescent; Children
MeSH Terms: conditions — Gambling; Internet Addiction Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaps prevention treatment (Experimental): The treatment will be administered in an individual format and consist of seven to nine sessions of 45 minutes over a period of seven to nine weeks. The number of sessions can vary to be able to accommodate the fact that participants may have different levels of motivation for changing their primary problem behavior, which is why some participants may require one or two extra sessions at the start of the treatment. The treatment will be offered to participants both in person and via video link to facilitate participation for children and adolescents living further away from the participating clinics.
  Interventions: Behavioral: Relaps Preventions Therapy
- Treatment as usual (Other): The patients in this arm will get treatment as usual at their Child and Adolescent psychiatry clinic.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Relaps Preventions Therapy — The treatment consists of three parts: 1) setting goals, 2) understanding and identifying high-risk situations and problem behaviors, and 3) consolidating the new activity schedule and identifying future high-risk behaviors. The first part is focused on examining the patient's undesirable behavior, his/her motivation for change, and establishing goals with the. The second part, drawing more from traditional Cognitive Behavioral Therapy (CBT) techniques, consists of exploring problematic situations, identifying high-risk situations and events, emotions and cognitions that induce the problematic gaming behavior or result in a relapse; managing game time with activity scheduling and practicing problem-solving skills. The final part consists of recognizing early warning signals that may indicate that the primary problem behavior is more likely to occur and consolidating the parts of the treatment that have been most helpful in maintaining the new activity schedule.
  Arms: Relaps prevention treatment
Behavioral: Treatment as usual — This group will receive treatment as usual at their Child and Adolescent Psychiatry Clinic.
  Arms: Treatment as usual

SUMMARY:
The aim of the study is twofold: 1) to evaluate an Relaps Prevention(RP) treatment for Problematic Gaming (PG) and Internet Gaming Disorder (IGD) patients recruited from child and youth psychiatry (CAP) clinics and 2) to test whether the quality of parent-child relationships plays role in the effect of RP treatment and vice versa - whether the RP treatment has a spillover effect on the quality of parent-child relationships.

DETAILED DESCRIPTION:
This study is a two-arm, parallel-group, single-blind, early-stage Randomized Clinical Trial (RCT) with embedded qualitative components. Participants will be randomized in a 1:1 ratio to either intervention or control, with a total of 162 participants (81+81) in the trial. The primary outcomes are measures of gaming and gambling behavior pre- and post-intervention, and the secondary outcomes include child ratings of parent-child communication, including parental knowledge, control and solicitousness about child gaming, as well as child disclosure and secrecy related to gaming.

Preliminary analyses will be conducted with regression analyses, paired sample t-tests and ANOVAs and performed in Mplus. In addition to the RCT, the study will be supplemented with a qualitative component with semi-structured individual interviews to capture participants' and clinicians' experiences of the treatment, as well as attitudes about parent-child relationships and parenting needs in carers whose children completed the RP treatment. The qualitative data will be analyzed with thematic analysis.

ELIGIBILITY:
Inclusion criteria

* age 12-18
* over cut-off on GASA
* over cut-off on CLiP

Exclusion criteria

* not being able to speak Swedish

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Gaming changes | treatment and 3 months
  Changes in gaming measured with Game Addiction Scale for Adolescents (GASA) . GASA applies to gaming behavior during the last 6 months with 7 items. Each question covers one criterion in the Diagnostic and Statistical Manual 5 (DSM-5), answered on a 5-point Likert scale ranging from 1 (never) to 5 (very often) and should according to the developer be counted as endorsed when rated 3 or higher.
  Min: 0 Max: 35 A higher outcome means worse gaming problems
Gambling changes | treatment and 3 months
  Changes in gambling measured with National Opinion Research Center (NORC) Diagnostic Screen for Gambling Disorders (NODS), three NODS questions, pertaining to loss of Control, Lying, and Preoccupation (CLiP).
  NODS-CLiP is the shorter form of NODS.
  Min: 0 Max:3 A higher outcome means worse gambling problems.

SECONDARY OUTCOMES:
Family climate/communication | treatment and 3 months
  Changes in family climate/communication.
  Parent-child communication includes six subscales. Items are rated on a five-point Likert scale ranging from 1 (often) to 5 (Never).
  Min: 0 Max: 30 A higher outcome means worse communication.
  Family climate , includes two subscales, family cohesion and conflict. While family cohesion assesses the bonds between family members, family conflict assesses the conflicts between family members. A total of 11 questions.
  Items are rated on a four-point scale, ranging from 1 (not true at all) to 4 (very true).
  Min: 0 Max: 44 A higher outcome means worse family climate.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Claesdotter-Knutsson, MD;PhD, Principal Investigator — emma.claesdotter-knutsson@skane.se
Locations (1):
- Child and adolescent Clinic Rehion Skane, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andre F, Kapetanovic S, Einarsson I, Trebbin Harvard S, Franzen L, Mottus A, Hakansson A, Claesdotter-Knutsson E. Relapse prevention therapy for internet gaming disorder in Swedish child and adolescent psychiatric clinics: a randomized controlled trial. Front Psychiatry. 2023 Oct 20;14:1256413. doi: 10.3389/fpsyt.2023.1256413. eCollection 2023. PMID 37928925
- [Derived] Kapetanovic S, Gurdal S, Einarsson I, Werner M, Andre F, Hakansson A, Claesdotter-Knutsson E. Relapse Prevention Therapy for Problem Gaming or Internet Gaming Disorder in Swedish Child and Youth Psychiatric Clinics: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 5;12:e44318. doi: 10.2196/44318. PMID 36602846